CLINICAL TRIAL: NCT01698567
Title: Antithrombin III Supplementation for Infants Undergoing Cardiac Surgery With Cardiopulmonary Bypass.
Brief Title: Antithrombin III in Infants With Cardiopulmonary Bypass (CPB)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Challenges enrolling subjects in study
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michael Eaton, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38402
Record Dates: First submitted 2012-09-04; First posted 2012-10-03 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Congenital Heart Disease
Keywords: Infants; Cardiopulmonary bypass; anticoaglution
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Antithrombin III; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antithrombin III (Active Comparator): Product- Antithrombin III is derived from pooled human plasma
  ATIII will be dosed using the formula recommended by the manufacturer:
  (goal activity - baseline activity) x weight (kg) x .714 (Assume: start with 35% activity [7], goal 120% activity[18], so dose = 120-35 x wt (kg) x .714, e.g. 5 kg infant: 85 x 5 x .714 = 303 units)
  a.
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator): placebo (normal saline)
  Interventions: Drug: Antithrombin III

INTERVENTIONS:
Drug: Antithrombin III — ATIII will be dosed using the formula recommended by the manufacturer:
  (goal activity - baseline activity) x weight (kg) x .714 (Assume: start with 35% activity [7], goal 120% activity[18], so dose = 120-35 x wt (kg) x .714, e.g. 5 kg infant: 85 x 5 x .714 = 303 units)
  Other Names: Thrombate
  Arms: Placebo
Drug: Placebo — placebo (normal saline) after induction of anesthesia and before commencement of bypass. ATIII will be dosed using the formula recommended by the manufacturer: (goal activity - baseline activity) x weight (kg) x .714 (Assume: start with 35% activity [7], goal 120% activity[18], so dose = 120-35 x wt (kg) x .714, e.g. 5 kg infant: 85 x 5 x .714 = 303 units)
  Other Names: Normal Saline
  Arms: Antithrombin III

SUMMARY:
The purpose of this study is to discern whether supplementation of Antithrombin III will decrease coagulation and inflammation associated with cardiopulmonary bypass in infants undergoing cardiac surgery.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) and cardiovascular surgery initiate diffuse activation of coagulation, inflammation and fibrinolysis that often has deleterious effects on patient outcomes, including bleeding, transfusion, myocardial dysfunction, renal failure, pulmonary dysfunction, prolonged intubation, ICU and hospital length of stay, stroke and neurocognitive dysfunction, and mortality.Pediatric patients are especially at risk for hematologic derangement related to CPB. Not only are infants and children subject to the same diffuse activations of coagulation, inflammation, and fibrinolysis as adults, but their size, immaturity, and circulatory abnormalities secondary to congenital heart disease increase the risk of loss of hematologic homeostasis. Since an infant's blood volume is much smaller than that of the prime in the CPB pump, hemodilution alone produces impaired hemostasis related to thrombocytopenia and coagulation factor dilution The incidence of each of these complications is variable and depends on the diagnosis, operation, time on CPB and other factors.

Adequate anticoagulation during cardiopulmonary bypass (CPB) is essential to preserve the hemostatic system and ensure hemostasis after surgery. Heparin has long been the mainstay of anticoagulation for CPB, due to its ease of use, familiarity, and reversibility. For heparin to exert its anticoagulant effect, it must bind with an intrinsic cofactor, antithrombin III (ATIII) to inhibit enzymes of the intrinsic and final common coagulation pathways. It has been established that neonates have significantly decreased levels of ATIII relative to adults, and that this relative deficiency continues at least until 6 months of age. Children with congenital heart disease have further decreases in ATIII and other abnormalities of coagulation which may contribute to adverse outcomes. Given this ATIII deficiency, it is not surprising that heparin anticoagulation does not fully suppress coagulation during CPB. Neonates anticoagulated for CPB with heparin have ongoing activation of humoral and cellular coagulation with associated activation of inflammation and fibrinolysis. Improved anticoagulation may reduce activation of these cascades and improve outcomes. In addition, infants are at high risk for post cardiac surgery intervascular thrombosis. Baseline ATIII deficiency, and consumption of ATIII during bypass may contribute to a postoperative prothrombotic state esulting in this often fatal complication. ATIII supplementation may decrease this risk.

ATIII is available as a lyophilized product derived from pooled human plasma. Treatment with ATIII has been shown to improve the anticoagulant effects of heparin and attenuate activation of hemostasis and inflammation during adult CPB, and to decrease the incidence of thrombosis associated with central venous cannulation in children. The incidence of central venous thrombosis in infants undergoing cardiac surgery has been reported as 5.8 - 22% in neonates, with a resultant mortality of 20%.

The biologic half-life of antithrombin in healthy adult volunteers is 2.5 - 3.8 days. Pharmacokinetic data in neonates is not available, but biologic activity should certainly persist through the 2 highest risk periods:

CPB, where activation of coagulation produces activation of inflammation, both cellular and humoral, and fibrinolysis.

The early post-op period when patients typically become hypercoagulable as part of the stress response to surgery. Hypercoagulability places the patients at high risk for central line-associated thrombosis despite by heparin-containing flush solutions which are standard of care. Ensuring a near normal level of antithrombin appears to enhance the ability of the flush solutions to inhibit thrombin generation on the catheter.

ATIII has been used in infants after cardiac surgery to prophylax against central venous thrombosis, for infants with necrotizing enterocolitis (NEC), and as treatment for neonates with congenital ATIII deficiency. Neonates appear to respond as expected to ATIII supplementation, with clinical efficacy for central venous thrombosis but not NEC. No complications unique to infants were reported in any of these publications.

It is reasonable to expect that ATIII would be even more beneficial in infants less than 6 months old.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included if they are presenting for elective cardiac surgery using cardiopulmonary bypass and are 180 days of age or less.

Exclusion Criteria:

Sensitivity to ATIII product (Thrombate, Grifols, Los Angeles, CA)

* Known inherited or acquired coagulation defect
* Current or prior treatment with pro-or anticoagulant medication within past 30 days (except aspirin or a single dose of heparin, e.g. for catheterization)
* Known central venous thrombosis
* Recent (30 days) transfusion with hemostatic blood products (fresh-frozen plasma, platelets, cryoprecipitate, whole blood)
* wt less than 3000g

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The primary hypothesis is that treatment with ATIII before bypass will decrease the activation of inflammation during CPB as measured by plasma neutrophil elastase. | Expected average of 24 months
  Patients treated with ATIII as standard of care (good clinical practice) will remain in the study and be analyzed by their intention to treat group. Review of our clinical experience shows that treatment with ATIII for heparin resistance occurs in 2-3% of cases. If there are more than two patients so treated, we will also perform an "as-treated" analysis.

SECONDARY OUTCOMES:
p-selectin | expected average of 24 months
interleukin-6 | Expected average of 24 months
prothrombin fragment 1.2 | expected average of 24 months
24 hour blood loss | 24 hours post surgery
ICU length of stay | Expected average of 3 days
Hospital length of stay | Expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eaton, MD, Principal Investigator — University of Rochester
Locations (1):
- Michael Eaton, MD, Rochester, New York, United States